CLINICAL TRIAL: NCT00251693
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of TAK-390MR (60 mg Once- Daily [QD] and 90 mg QD) and an Active Comparator, Lansoprazole (30 mg QD) on Healing of Erosive Esophagitis
Brief Title: Efficacy and Safety of Dexlansoprazole MR and Lansoprazole on Healing of Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T-EE04-084; U1111-1113-9373 (Registry Identifier: WHO)
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Results first posted 2009-03-23 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Esophagitis, Reflux; Esophagitis, Peptic
Keywords: Erosive Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexlansoprazole MR 60 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Dexlansoprazole MR 90 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Lansoprazole 30 mg QD (Active Comparator)
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole MR — Dexlansoprazole MR 60 mg, capsules, orally, once daily (QD) for up to 8 weeks.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 60 mg QD
Drug: Dexlansoprazole MR — Dexlansoprazole MR 90 mg, capsules, orally, once daily for up to 8 weeks.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 90 mg QD
Drug: Lansoprazole — Lansoprazole 30 mg, capsules, orally, once daily for up to 8 weeks.
  Other Names: Prevacid; AG-1749
  Arms: Lansoprazole 30 mg QD

SUMMARY:
The purpose of this study is to assess the efficacy and safety of 8 weeks of once-daily (QD) treatment with dexlansoprazole modified release (MR) 60 mg or 90 mg or lansoprazole 30 mg in healing subjects with endoscopically proven erosive esophagitis.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, multi-center, active-controlled, 3-arm study with an 8-week treatment period. This study will compare the efficacy of dexlansoprazole MR (60 mg QD and 90 mg QD) with that of lansoprazole (30 mg) when administered orally as a single daily dose in the morning, before breakfast. The study is designed to evaluate healing of erosive esophagitis and the effect of the therapy on relieving gastroesophageal reflux disease-related symptoms. The study consists of two periods, a screening period (maximum 21 days) and a treatment period, which will last 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have endoscopically confirmed erosive esophagitis as defined by the Los Angeles (LA) Classification Grading System (A-D)

Exclusion Criteria:

* Subject has a positive Campylobacter-like organisms (CLO) test for Helicobacter (H.) pylori.
* Use of prescription or non-prescription proton pump inhibitors (PPIs), histamine (H2) receptor antagonists or sucralfate, drugs with significant anticholinergic effects, misoprostol or prokinetics
* Use of antacids [except for study supplied Gelusil®]
* Need for continuous anticoagulant therapy (blood thinners)
* Endoscopic Barrett's esophagus and/or definite dysplastic changes in the esophagus
* History of dilatation of esophageal strictures, other than Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter)
* Current or historical evidence of Zollinger-Ellison syndrome or other hypersecretory condition.
* History of gastric, duodenal or esophageal surgery except simple oversew of an ulcer.
* Acute upper gastrointestinal hemorrhage within 4 weeks of the screening endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2038 (Actual)
Dates: Start 2005-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda
Locations (140):
- United States (96):
  - Alabaster, Alabama
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Chula Vista, California
  - Fullerton, California
  - Garden Grove, California
  - Irvine, California
  - Lancaster, California
  - Long Beach, California
  - Los Angeles, California
  - Mission Hills, California
  - Palm Springs, California
  - Pasadena, California
  - Redwood City, California
  - San Diego, California
  - San Luis Obispo, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Lone Tree, Colorado
  - Wheat Ridge, Colorado
  - Waterbury, Connecticut
  - Boynton Beach, Florida
  - Jacksonsville, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Lakeland, Florida
  - New Port Richey, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Hines, Illinois
  - Oak Park, Illinois
  - Rockford, Illinois
  - Clive, Iowa
  - Dubuque, Iowa
  - Newton, Kansas
  - Shawnee Mission, Kansas
  - Topeka, Kansas
  - Metairie, Louisiana
  - Shreveport, Louisiana
  - Hollywood, Maryland
  - Lutherville, Maryland
  - Troy, Michigan
  - Chaska, Minnesota
  - Jackson, Mississippi
  - Mexico, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Omaha, Nebraska
  - Pahrump, Nevada
  - Binghamton, New York
  - Brooklyn, New York
  - Great Neck, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Elkin, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Mayfield Heights, Ohio
  - Warren, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Beaver Falls, Pennsylvania
  - Duncansville, Pennsylvania
  - Lansdale, Pennsylvania
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Hermitage, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Beaumont, Texas
  - Byran, Texas
  - Corsicana, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Ogden, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Chesapeake, Virginia
  - Danville, Virginia
  - Spokane, Washington
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin
- Australia (2):
  - Box Hill
  - South Brisbane
- Sofia, Bulgaria
- Canada (6):
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Québec, Quebec
  - Regina, Saskatchewan
  - Saskatoon, Saskatchewan
- Prague, Czechia
- Germany (4):
  - Hamburg, Hamburg
  - Dietzenback, Hesse
  - Schweim, North Rhine-Westphalia
  - Borna, Saxony
- Gyula, Hungary
- India (10):
  - Gujarat, Ahmedabad
  - Tamilnadu, Chennai
  - Rajasthan, Jaipur
  - Ludhiana, Punjab
  - Madurai, Tamina
  - Chennai
  - Coimbatore
  - Hyderabad
  - New Delhi
  - Visakhapatnam
- Riga, Latvia
- Kaunas, Lithuania
- Hamilton, New Zealand
- Lima, Peru
- Poland (4):
  - Krakow
  - Lubin
  - Sopot
  - Warzawa
- Slovakia (4):
  - Bratislava
  - Nitra
  - Sučany
  - Tmava
- South Africa (7):
  - Gauteng, Johannesburg
  - Cape Town, WC
  - Panorama, WC
  - Pinelands, WC
  - Plumstead, WC
  - Somerset West, WC
  - Pretoria

REFERENCES:
- [Result] Sharma P, Shaheen NJ, Perez MC, Pilmer BL, Lee M, Atkinson SN, Peura D. Clinical trials: healing of erosive oesophagitis with dexlansoprazole MR, a proton pump inhibitor with a novel dual delayed-release formulation--results from two randomized controlled studies. Aliment Pharmacol Ther. 2009 Apr 1;29(7):731-41. doi: 10.1111/j.1365-2036.2009.03933.x. PMID 19183157
- [Result] Peura DA, Metz DC, Dabholkar AH, Paris MM, Yu P, Atkinson SN. Safety profile of dexlansoprazole MR, a proton pump inhibitor with a novel dual delayed release formulation: global clinical trial experience. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1010-21. doi: 10.1111/j.1365-2036.2009.04137.x. Epub 2009 Sep 4. PMID 19735233
- [Result] Wyrwich KW, Mody R, Larsen LM, Lee M, Harnam N, Revicki DA. Validation of the PAGI-SYM and PAGI-QOL among healing and maintenance of erosive esophagitis clinical trial participants. Qual Life Res. 2010 May;19(4):551-64. doi: 10.1007/s11136-010-9620-x. Epub 2010 Feb 27. PMID 20195905
- [Result] Friedlander EA, Pallentino J, Miller SK, VanBeuge SS. The evolution of proton pump inhibitors for the treatment of gastroesophageal reflux disease. J Am Acad Nurse Pract. 2010 Dec;22(12):674-83. doi: 10.1111/j.1745-7599.2010.00578.x. Epub 2010 Nov 24. PMID 21129076
- [Derived] Peura DA, Pilmer B, Hunt B, Mody R, Perez MC. Distinguishing the impact of dexlansoprazole on heartburn vs. regurgitation in patients with gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2013 Nov;38(10):1303-11. doi: 10.1111/apt.12504. Epub 2013 Sep 30. PMID 24118079
- [Derived] Peura DA, Pilmer B, Hunt B, Mody R, Perez MC. The effects of increasing body mass index on heartburn severity, frequency and response to treatment with dexlansoprazole or lansoprazole. Aliment Pharmacol Ther. 2013 Apr;37(8):810-8. doi: 10.1111/apt.12270. Epub 2013 Mar 4. PMID 23451835
- See also: For the Dexilant Package Insert refer to this link — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 95 sites in the United States (US) and 55 ex-US sites from 02 December 2005 to 30 January 2007.
Pre-assignment Details: Subjects recorded day and nighttime heartburn symptoms and rescue medications for a screening period of up to 21 days. Subjects with endoscopically-proven erosive esophagitis (EE) at screening were enrolled in Dexlansoprazole Modified Release (MR) or Lansoprazole once daily (QD) treatment group.
Groups:
- Dexlansoprazole MR 60 mg QD: Dexlansoprazole MR 60 mg, capsules, orally, once daily for up to 8 weeks.
- Dexlansoprazole MR 90 mg QD: Dexlansoprazole MR 90 mg, capsules, orally, once daily for up to 8 weeks.
- Lansoprazole 30 mg QD: Lansoprazole 30 mg, capsules, orally, once daily for up to 8 weeks.
Period: Overall Study
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Lansoprazole 30 mg QD
Started | 680 | 668 | 690
Completed | 629 | 624 | 644
Not Completed | 51 | 44 | 46
Not completed — Adverse Event | 17 | 9 | 9
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Lost to Follow-up | 12 | 7 | 8
Not completed — Withdrawal by Subject | 11 | 17 | 14
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Inclusion/exclusion criteria not met | 5 | 3 | 8
Not completed — Noncompliant | 0 | 0 | 2
Not completed — Possible Barrett's esophagus | 3 | 5 | 2
Not completed — Subject request/subject unavailable | 1 | 2 | 0
Not completed — Abnormal laboratory findings | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Lansoprazole 30 mg QD | Total
Number analyzed (Participants) | 680 | 668 | 690 | 2038
Age, Customized [Number; unit: participants]
  <45 Years | 269 | 276 | 288 | 833
  45 Years to <65 Years | 349 | 328 | 332 | 1009
  >=65 Years | 62 | 64 | 70 | 196
Age Continuous [Mean (Standard Deviation); unit: years] | 47.8 (13.71) | 47.3 (13.93) | 47.3 (13.74) | 47.5 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300 | 302 | 325 | 927
  Male | 380 | 366 | 365 | 1111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 52 | 54 | 166
  Not Hispanic or Latino | 620 | 616 | 636 | 1872
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 4 | 7 | 17
  Asian | 27 | 33 | 33 | 93
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 32 | 33 | 27 | 92
  White | 602 | 580 | 601 | 1783
  More than one race | 10 | 15 | 17 | 42
  Unknown or Not Reported | 2 | 3 | 4 | 9
Los Angeles (LA) Classification Grade for Erosive Esophagitis (EE) [Number; unit: Paricipants] — LA Classification for Esophagitis Grading System (grades A, B, C, D) with increasing severity from grade A to grade D.
  Paricipants
    A: ≥1 mucosal break <5mm | 236 | 242 | 231 | 709
    B: ≥1 mucosal break ≥5mm | 247 | 233 | 248 | 728
    C: ≥1 mucosal break and <75% of the circumference | 163 | 148 | 170 | 481
    D: ≥1 mucosal break and ≥75% of the circumference | 33 | 45 | 40 | 118
    Not Applicable | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Complete Healing of Erosive Esophagitis (EE) by Week 8 as Assessed by Endoscopy - Crude Rate Analysis.
Description: Percentage of subjects with complete healing of EE as assessed by endoscopy was analyzed for change in LA Esophagitis Classification grades A, B, C, or D to healed. Healed is defined as anything that is less than the criterion for Grade A (greater than or equal to 1 mucosal break and less than 5 mm). If it doesn't meet the A criterion, it's counted as healed.
Time Frame: 8 Weeks
Population: Crude rate analyses were performed on the ITT subjects who had at least 1 post-baseline endoscopy assessment performed within 7 days of the last day of study drug.
Measure: Number; unit: Percentage of subjects
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Lansoprazole 30 mg QD
Number analyzed (Participants) | 639 | 634 | 656
Percentage of subjects | 85.3 [82.3 to 87.9] | 85.8 [82.8 to 88.4] | 79.0 [75.6 to 82.0]
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Lansoprazole 30 mg QD; Test type: Non-Inferiority or Equivalence — If the lower bound of the 95% CI was greater than -10%, noninferiority was concluded. Superiority of primary efficacy endpoint was assessed by comparing the crude healing rate of dexlansoprazole MR 60 mg dose to that of lansoprazole 30 mg using a Cochran Mantel Haenszel (CMH) test with baseline LA EE Grade as strata; p = 0.004, Cochran-Mantel-Haenszel — Unadjusted p-value is presented. The overall 0.05 level of significance for the multiple comparisons of each dexlansoprazole dose to lansoprazole was controlled using Hochberg's method; Difference in percentage = 6.33, 95% CI [2.17 to 10.48]
Statistical Analysis 2: Comparison: Dexlansoprazole MR 90 mg QD vs Lansoprazole 30 mg QD; Test type: Non-Inferiority or Equivalence — If the lower bound of the 95% CI was greater than -10%, noninferiority was concluded. Superiority of primary efficacy endpoint was assessed by comparing the crude healing rate of dexlansoprazole MR 90 mg dose to that of lansoprazole 30 mg using a Cochran Mantel Haenszel (CMH) test with baseline LA EE Grade as strata; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 6.84, 95% CI [2.70 to 10.98]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.727, Cochran-Mantel-Haenszel — Statistical significance was determined at the 0.05 level without adjustment for multiple comparisons

2. Secondary Outcome: Percentage of Subjects With Baseline Erosive Esophagitis Grade C or D Combined Who Have Complete Healing of Erosive Esophagitis by Week 8 as Assessed by Endoscopy - Crude Rate Analysis.
Description: Percentage of subjects with baseline EE grade C or D combined who have complete healing of erosive esophagitis as assessed by endoscopy for Change in LA Esophagitis Classification Grades C and D to healed. Healed is defined as anything that is less than the criterion for Grade A. If it doesn't meet the A criterion, it's counted as healed.
Time Frame: 8 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Lansoprazole 30 mg QD
Number analyzed (Participants) | 182 | 185 | 200
percentage of subjects | 79.7 [73.1 to 85.3] | 74.1 [67.1 to 80.2] | 65.0 [58.0 to 71.6]
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Lansoprazole 30 mg QD; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — Unadjusted p-value is presented. Statistical significance was determined at 0.05 level by Hommel-Simes method within treatment and Hochberg method for comparisons of each dexlansoprazole dose to lansoprazole
Statistical Analysis 2: Comparison: Dexlansoprazole MR 90 mg QD vs Lansoprazole 30 mg QD; Test type: Superiority or Other; p = 0.045, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.245, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

3. Secondary Outcome: Percentage of Subjects With Baseline Erosive Esophagitis Grade C or D Combined Who Have Complete Healing of Erosive Esophagitis by Week 8 as Assessed by Endoscopy - Life Table Method.
Description: Percentage of subjects with baseline EE grade C or D combined who have complete healing of EE as assessed by endoscopy for Change in LA Esophagitis Classification Grades C and D to healed. Healed is defined as anything that is less than the criterion for Grade A. If it doesn't meet the A criterion, it's counted as healed.
Time Frame: 8 Weeks
Population: In addition to the ITT subjects who had at least 1 post-baseline endoscopy, Life Table Method included the ITT subjects without any post-baseline endoscopy within 7 days of the last day of study drug as censored.
Measure: Number; unit: percentage of subjects
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Lansoprazole 30 mg QD
Number analyzed (Participants) | 191 | 191 | 208
percentage of subjects | 88.9 [83.7 to 94.2] | 83.8 [77.4 to 90.1] | 74.5 [67.3 to 81.6]
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Lansoprazole 30 mg QD; Test type: Superiority or Other; p = 0.011, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Dexlansoprazole MR 90 mg QD vs Lansoprazole 30 mg QD; Test type: Superiority or Other; p = 0.017, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.927, Log Rank — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

4. Primary Outcome: Percentage of Subjects With Complete Healing of Erosive Esophagitis by Week 8 as Assessed by Endoscopy - Life Table Method.
Description: Percentage of subjects with complete healing of EE as assessed by endoscopy was analyzed for change in LA Esophagitis Classification grades A, B, C, or D to healed. Healed is defined as anything that is less than the criterion for Grade A. If it doesn't meet the A criterion, it's counted as healed.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Lansoprazole 30 mg QD
Number analyzed (Participants) | 673 | 665 | 684
Percentage of subjects | 92.3 [90.0 to 94.7] | 92.2 [89.8 to 94.6] | 86.1 [83.0 to 89.2]
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Lansoprazole 30 mg QD; Test type: Non-Inferiority or Equivalence — Noninferiority was supported if the lower bound of the 95% CI for the difference with lansoprazole 30 mg of the estimated 8-week healing rate was greater than -10%. Superiority was assessed based on log-rank tests comparing treatments for the endpoints; p = 0.060, Log Rank — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 6.20, 95% CI [2.30 to 10.11]
Statistical Analysis 2: Comparison: Dexlansoprazole MR 90 mg QD vs Lansoprazole 30 mg QD; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.029, Log Rank — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = 6.08, 95% CI [2.16 to 10.00]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.707, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

5. Secondary Outcome: Percentage of Subjects With Complete Healing of Erosive Esophagitis by Week 4 as Assessed by Endoscopy - Crude Rate Analyses.
Description: as for outcome 4
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Lansoprazole 30 mg QD
Number analyzed (Participants) | 639 | 634 | 656
Percentage of subjects | 66.2 [62.4 to 69.9] | 68.8 [65.0 to 72.4] | 64.8 [61.0 to 68.4]
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Lansoprazole 30 mg QD; Test type: Superiority or Other; p = 0.705, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Dexlansoprazole MR 90 mg QD vs Lansoprazole 30 mg QD; Test type: Superiority or Other; p = 0.146, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.283, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

6. Secondary Outcome: Percentage of Subjects With Complete Healing of Erosive Esophagitis by Week 4 as Assessed by Endoscopy - Life Table Method.
Description: as for outcome 4
Time Frame: 4 Weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Lansoprazole 30 mg QD
Number analyzed (Participants) | 673 | 665 | 684
Percentage of subjects | 77.0 [73.5 to 80.5] | 78.8 [75.4 to 82.2] | 76.5 [73.0 to 80.0]
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Lansoprazole 30 mg QD; Test type: Superiority or Other; p = 0.896, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Dexlansoprazole MR 90 mg QD vs Lansoprazole 30 mg QD; Test type: Superiority or Other; p = 0.241, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.211, Log Rank — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

ADVERSE EVENTS:
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Lansoprazole 30 mg QD
Serious Adverse Events (participants affected / at risk) | 5/680 | 2/668 | 6/690
Other Adverse Events (participants affected / at risk) | 63/680 | 53/668 | 50/690
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole MR 60 mg QD (N=680) | Dexlansoprazole MR 90 mg QD (N=668) | Lansoprazole 30 mg QD (N=690)
Coronary Artery Disorders not elsewhere classified (NEC) (Cardiac disorders) | 1 | 0 | 0
Duodenal and Small Intestinal Stenosis and Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal (GI) Atonic and Hypomotility Disorders NEC (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Inflammatory Disorders NEC (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids and GI Varices (Excluding [Excl] Oesophageal) (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Ulcers and Perforation NEC (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal and Retroperitoneal Disorders (Gastrointestinal disorders) | 1 | 0 | 0
Pain and Discomfort NEC (General disorders) | 1 | 0 | 0
Cholecystitis and Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Infections NEC (Infections and infestations) | 1 | 0 | 0
Lower Respiratory Tract and Lung Infections (Infections and infestations) | 1 | 0 | 0
Sepsis, Bacteraemia, Viraemia and Fungaemia NEC (Infections and infestations) | 1 | 0 | 0
Streptococcal Infections (Infections and infestations) | 0 | 0 | 1
Non-site Specfic Procedural Complications (Injury, poisoning and procedural complications) | 0 | 0 | 1
Potassium Imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Soft Tissue Disorders NEC (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute Polyneuropathies (Nervous system disorders) | 1 | 0 | 0
Transient Cerebrovascular (CV) Events (Nervous system disorders) | 1 | 0 | 0
Paralysis and Paresis (Excl Cranial Nerve) (Nervous system disorders) | 0 | 0 | 1
Central Nervous System Hemorrhages and CV accidents (Nervous system disorders) | 0 | 0 | 1
Bipolar Disorders (Psychiatric disorders) | 0 | 0 | 1
Respiratory Failures (Excl Neonatal) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole MR 60 mg QD (N=680) | Dexlansoprazole MR 90 mg QD (N=668) | Lansoprazole 30 mg QD (N=690)
Diarrhoea (Excl Infective) (Gastrointestinal disorders) | 27 | 24 | 21
Gastrointestinal and Abdominal Pains (Excl Oral and Throat) (Gastrointestinal disorders) | 17 | 24 | 17
Upper Respiratory Tract Infections (Infections and infestations) | 24 | 17 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.